CLINICAL TRIAL: NCT06759064
Title: Efficacy and Safety of Intraperitoneal Immune Checkpoint Inhibitors and Zoledronic Acids in Gastric Cancer Malignant Ascites: a Phase I/II Clinical Study (IPIZA)
Brief Title: Intraperitoneal Immune Checkpoint Inhibitors and Zoledronic Acids for Gastric Cancer Malignant Ascites
Acronym: IPIZA
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Lian Liu, MD, PHD, Professor, Qilu Hospital of Shandong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IPIZA
Record Dates: First submitted 2024-12-10; First posted 2025-01-06 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Cancer of Stomach, Adenocarcinoma; Ascites, Malignant
Keywords: gastric cancer; malignant ascites; Immune checkpoint inhibitors; zoledronic acid; intraperitoneal injection
MeSH Terms: conditions — Stomach Neoplasms; Adenocarcinoma; Ascites | interventions — Zoledronic Acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- zoledronic acid plus Sintilimab intraperitoneal injection therapy arm (Experimental): patients will receive zoledronic acid 0.5-1mg plus Sintilimab 1.0mg/kg intraperitoneal injection
  Interventions: Drug: zoledronic acid plus Sintilimab intraperitoneal injection

INTERVENTIONS:
Drug: zoledronic acid plus Sintilimab intraperitoneal injection — At D-5~D-1, drain the ascites by placing a tube in the abdominal cavity first, try to drain the ascites as much as possible according to the clinical routine, and record the amount of drainage.D1, D8, D15, D22 start the first immunocheckpoint inhibitor combined with zoledronic acid treatment, try to drain the ascites first, calculate the amount of drugs according to the patient's body weight, and then dissolve the corresponding dosage of immunocheckpoint inhibitor and zoledronic acid in 100 ml of saline and inject them into the abdominal cavity respectively, and then inject another 100 ml of saline according to the patient's tolerance. The corresponding dose of immune checkpoint inhibitor and zoledronic acid was dissolved in 100 ml of saline and injected into the abdominal cavity.

SUMMARY:
This study is to evaluate the safety and efficacy of intraperitoneal injection of immune checkpoint inhibitor combined with zoledronic acid for the treatment of malignant ascites in gastric cancer.

This study is a phase Ib/II clinical study to evaluate the safety and efficacy of intraperitoneal injection of immune checkpoint inhibitors in combination with zoledronic acid in the treatment of malignant ascites in gastric cancer, which consists of two phases, firstly, the phase Ib safety study, which adopts the '3+3' drug-escalation experimental design, and after determining the safe and tolerable dose, it will proceed to the second part of the phase II efficacy study. The Phase II study was designed by Simon's two-stage approach to evaluate the efficacy of immune checkpoint inhibitors in combination with zoledronic acid in the treatment of malignant ascites in gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* Gastric adenocarcinoma diagnosed pathologically;
* Malignant ascites confirmed by ascites cytology;
* Presence of ascites confirmed by CT with ascites graded as 2nd and 3rd degree (EASL guidelines and ICA consensus);
* Those aged 18-75 years;
* Patients who had not undergone local administration of drugs in the abdominal cavity and systemic immunotherapy within the previous 4 weeks;
* Vital signs are stable, Karnofsky score (≥70), and expected survival time is >3 months;
* Normal bone marrow haematopoietic function, blood routine: HGB ≥90g/L, WBC ≥2.5×10^9/L (NEU ≥1.5×10^9/L), PLT ≥90×10^9/L;
* Normal coagulation function without bleeding tendency (International normalised ratio of prothrombinogen INR<1.5);
* Liver function: total bilirubin ≤1.5 times the upper limit of normal (ULN); AST and ALT ≤2 times the upper limit of normal (ULN) (or ≤5 times the upper limit of normal (ULN) if the abnormalities are mainly due to tumour infiltration);
* Renal function: Cr ≤1.5 times the upper limit of normal (ULN) or creatinine clearance ≥60mL/min.

Exclusion Criteria:

* Non-malignant ascites (e.g., portal hypertension ascites or infected ascites);
* Presence of contraindications to immunotherapy (including long-term hormone use, history of radiation pneumonitis, radiation hepatitis, radiation enteritis, etc.);
* Combination of other serious cardiopulmonary diseases that affect the treatment, etc;
* Patients with extensive abdominal adhesions; encapsulated peritoneal fluid; history of intestinal obstruction; and malignant patients with extensive distant metastases in the terminal stage;
* Women who are breastfeeding, pregnant, or preparing for pregnancy;
* Patients with plasma albumin (ALB) <30 g/L and severe hypoproteinemia;
* Patients with known hypersensitivity to components of the test drug or its analogues;
* Patients with other severe, acute or chronic diseases that may interfere with the interpretation of the study results and who, in the judgement of the investigator, are unsuitable for participation in the clinical trial;
* Patients with cognitive dysfunction, or poor treatment compliance as judged by the investigator;
* Participants in other clinical trials within 4 weeks;
* Combination of other malignancies;
* Those who, in the opinion of the investigator, are not suitable for participation in the clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-09-12 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) or maximal tolerance dose (MTD) in the Phase Ib stage | 28 days after the last treatment
  Side effects of drug or treatment that are serious enough (e. g. ≥Grade 3 non-hematologic toxicity according to CTCAE 5.0 in ≥1/3) to prevent an increase in dose or level of that treatment. The MTD is defined as the previous dose level.
Objective response rate | 4 weeks after last treatment
  Complete remission (CR): complete resolution of ascites and maintained for more than 4 weeks; complete disappearance of all target lesions; Partial remission (PR): the amount of CT-measured ascites decreased by more than 50% compared to pretreatment and the amount of ascites withdrawn again was less than 1/2 of the previous withdrawal and was maintained for more than 4 weeks; the sum of the diameters of all measurable target lesions was ≥30% below baseline; Objective Response Rate（ORR） = CR + PR

SECONDARY OUTCOMES:
Rates of Adverse events according to CTCAE 5.0 in overall subjects | 3 months after the last treatment
  Adverse events were graded and recorded according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0. A general physical examination, measurement of vital signs, laboratory safety evaluation, and documentation of relevant adverse events were performed at each visit during the treatment period.
Time for ascites control | 1 year
  If PD was judged and ascites was not re-punctured and drained, the time of this follow-up visit was used as the time of ascites control; if the patient had undergone puncture and drainage prior to the follow-up visit due to intolerance of ascites symptoms, the time of re-puncture was used as the time of ascites control.
Immune cell changes | 4 weeks
  Immune cell changes in ascites
Quality of Life Assessment | 1 year
  A quality of life score (QOL) for oncology patients was used. The quality of life score (QOL) of oncology patients contains 12 dimensions, including appetite, spirit, sleep, fatigue, pain, family understanding and cooperation, colleagues' understanding and cooperation (including leadership), own knowledge of cancer, attitude towards treatment, daily life, side effects of treatment, and facial expression, with the highest score of 5 and the lowest score of 1 for each dimension. Quality of life grading: Quality of life is scored out of 60, with 51-60 for good, 41-50 for better, 31-40 for average, 21-30 for poor, and <20 for very poor quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No